CLINICAL TRIAL: NCT00440375
Title: Effects of Rosiglitazone on Bone in Postmenopausal Diabetic Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KA 05/74
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Menopause
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
The purpose of this study is to evaluate the effect of rosiglitazone on bone metabolism and to assess the association between the changes in bone turnover parameters and plasma cytokine levels in postmenopausal diabetic women

DETAILED DESCRIPTION:
Fifty-six obese, drug naive patients with type 2 diabetes mellitus were enrolled and completed the study. Twenty-six healthy subjects matched for age and body mass index (BMI) served as nondiabetic controls. All subjects were postmenopausal women with last menses at least 2 years. After the baseline measurements, all subjects were instructed to follow a weight-maintaining diet, based on ADA recommendations, and were also encouraged to walk or to jog at least 30 min daily. Subsequently, 28 of the diabetic subjects were randomly assigned to receive rosiglitazone (4 mg/day). Twenty-eight of diabetic subjects were on diet alone. The randomization procedure was based on a random sequence.

All subjects had a complete clinical examination, anthropometric measurements, and laboratory tests at baseline and at the end of the 12th week of the study. Laboratory investigations included assessment of: (i) glycemic control (HbA1c, fasting plasma glucose and insulin levels, and homeostasis model assessment (HOMA) index (22); (ii) serum bsALP and active human osteocalcin concentration (OCL) as markers of bone formation; (iii) urine deoxypyridinoline (DPD) as marker of bone resorption. Other non-specific bone markers including serum total ALP activity, urinary calcium (Ca) and phosphate (PO4) concentrations were also measured. Urine concentrations of DPD (nmol/L), Ca and PO4 (both in mmol/L) were corrected for their respective urine creatinine (Cr) concentrations in mmol/L (Urine DPD/Cr, Urine Ca/Cr and Urine PO4/Cr respectively). In addition, fasting blood samples were analyzed for plasma cytokine levels including IL-1β, IL-6 and TNF-α, and for haptoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes mellitus
* Postmenopausal period

Exclusion Criteria:

* Recent fracture or osteoporosis
* Drugs that may affect calcium or bone metabolism or drugs known to interfere with cytokine release
* Thyroid, parathyroid, pituitary, nutritional, inflammatory, hepatic, renal, or neoplastic disorders
* Severe cardiovascular disease

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82
Dates: Start 2005-06; Study Completion 2006-03

PRIMARY OUTCOMES:
metabolic bone markers before and after the intervention,

SECONDARY OUTCOMES:
association between the changes in bone turnover parameters and plasma cytokine levels

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Berberoglu, Principal Investigator — The Society of Endocrinology and Metabolism of Turkey

REFERENCES:
- [Derived] Berberoglu Z, Gursoy A, Bayraktar N, Yazici AC, Bascil Tutuncu N, Guvener Demirag N. Rosiglitazone decreases serum bone-specific alkaline phosphatase activity in postmenopausal diabetic women. J Clin Endocrinol Metab. 2007 Sep;92(9):3523-30. doi: 10.1210/jc.2007-0431. Epub 2007 Jun 26. PMID 17595249